CLINICAL TRIAL: NCT00076986
Title: PRECISE - Phase III Randomized Evaluation of Convection Enhanced Delivery of IL13-PE38QQR Compared to GLIADEL® Wafer With Survival Endpoint in Glioblastoma Multiforme Patients at First Recurrence
Brief Title: The PRECISE Trial: Study of IL13-PE38QQR Compared to GLIADEL Wafer in Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IL13PEI-301-R03; PRECISE Trial; NCT00090948 (obsolete NCT alias)
Record Dates: First submitted 2004-02-06; First posted 2004-02-10 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Glioblastoma Multiforme
Keywords: brain tumor; recurrent malignant glioma; brain neoplasm; central nervous system; surgery; resection; GLIADEL; infusion; glioblastoma multiforme; convection-enhanced delivery; first recurrence; recurrent GBM; GBM; supratentorial GBM
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma | interventions — IL13-PE38; Surgical Procedures, Operative; Carmustine

INTERVENTIONS:
Drug: IL13-PE38QQR
Procedure: surgery and catheter placement (2 procedures)
Drug: prolifespan 20 with carmustine implant (GLIADEL® Wafer)
Procedure: surgery and wafer placement (1 procedure)

SUMMARY:
The purpose of the PRECISE trial is to determine whether overall survival duration, safety, and quality of life are improved for patients treated with IL13-PE38QQR compared to patients treated with GLIADEL® Wafer following surgical tumor removal in the treatment of first recurrence of glioblastoma multiforme.

DETAILED DESCRIPTION:
PRECISE is a Phase III clinical trial of experimental drug IL13-PE38QQR (Study Drug). IL13-PE38QQR is a tumor-targeting agent administered by a continuous infusion directly into the brain around the cavity where the tumor has been removed. Through previous research, this Study Drug has shown potential to control some of the recurrent malignant gliomas, such as glioblastoma multiforme (GBM), anaplastic astrocytoma, and malignant mixed oligoastrocytoma.

The Study Drug is made by combining a human protein (IL13) with a portion of a bacterial toxin protein, Pseudomonas Exotoxin (PE). The IL13 portion binds to receptors on the tumor like a "key to a lock," allowing the PE portion to enter and kill those cells. Since tumor cells preferentially bind the drug, normal (healthy) brain cells are much less likely to be damaged by the drug. The Study Drug is delivered through tubing or catheters placed directly into the area surrounding the resection cavity. These catheters will be surgically placed from 2-7 days after the tumor has been removed. A pump is then used to slowly push the drug solution through the catheters using convection-enhanced delivery (CED) over a period of 4 days.

The GLIADEL® Wafer is an anti-cancer drug that is approved by the U.S. Food and Drug Administration (FDA) and sold for the treatment of recurrent or newly diagnosed GBM. Patients receiving GLIADEL® will have wafers placed at the time of surgery to remove tumor.

Eligible patients enrolled in the PRECISE trial will be randomly assigned to receive either IL13-PE38QQR or GLIADEL® Wafer. Patients will have a 2 out of 3 chance to receive IL13-PE38QQR and 1 out of 3 chance to receive GLIADEL® Wafer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old.
* Patients must have clinical and/or radiographic evidence of FIRST recurrence or progression of supratentorial GBM afer a previous resection or biopsy and external beam radiation therapy.
* Patients must have histopathologic documentation of GBM at initial diagnosis.
* Patients must have had previous cytoreductive surgery or biopsy for GBM.
* Patients must have received external beam radiotherapy with ≥ 45 Gy tumor dose, completed ≥ 4 weeks prior to study entry.
* Gross total resection (i.e., ≥ 95% resection of the solid, contrast-enhancing tumor component) must be planned.
* Tumor must have a solid contrast-enhancing component ≥ 1.0 cm in diameter. Baseline measurements must be obtained ≤ 2 weeks prior to study entry.
* Patients must be in adequate condition, as indicated by:

  1. Karnofsky Performance Score ≥ 70,
  2. Adequate hematologic status: i. Absolute neutrophil count (ANC) ≥ 1,500/mm3; ii. Hemoglobin ≥ 10 gm/dL; iii. Platelets ≥ 100,000/mm3; iv. PT and aPTT ≤ 1.5 x institutional upper limit
* Patients must not be receiving concurrent anti-tumor therapy and must have recovered from toxicity of prior therapy. Minimum intervals required:
* ≥ 6 weeks after receiving nitrosourea cytotoxic drug
* ≥ 4 weeks after receiving any non-nitrosourea cytotoxic drug or any systemic investigational agent
* ≥ 2 weeks after receiving any non-cytotoxic anti-tumor drug (including celecoxib or other drugs, if they are being used as anti-tumor therapies)
* Patients must be willing to practice an effective method of birth control during the study. Female patients must not be pregnant or breast-feeding.
* Patients or legal representative must understand the investigational nature of this study and sign a written informed consent form, approved by an Institutional Review Board (IRB) or an Independent Ethics Committee (IEC), prior to performance of any study-specific procedure

Exclusion Criteria:

* Patients with contrast-enhancing tumor component crossing the midline, multi-focal tumor not amenable to gross total resection, or tumor dissemination (subependymal or leptomeningeal).
* Expected communication between ventricle and resection cavity that cannot be repaired in order to safely use GLIADEL® Wafer.
* Patients with clinically significant increased intracranial pressure (e.g., impending herniation), uncontrolled seizures, or requirement for immediate palliative treatment.
* Patients who have received any type of stereotactic radiosurgery or brachytherapy, with the exception of the stereotactic radiosurgery boost part of the initial fractionated external beam radiation therapy.
* Patients who have received:

  1) prior treatment with IL13-PE38QQR, or, 2) GLIADEL® Wafer, or, 3) any intracerebral investigational agent
* Patients who have demonstrated a previous hypersensitivity to BCNU or any other component of the GLIADEL® Wafer.
* Patients unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (40):
  - University of Alabama at Birmingham - Division of Neurosurgery, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Los Angeles County/USC, Los Angeles, California
  - Cedars-Sinai Medical Center - Neurological Institute, Los Angeles, California
  - University of California - Los Angeles Neuro-Oncology Program, Los Angeles, California
  - University of California San Francisco - Dept. of Neurological Surgery, San Francisco, California
  - University of Colorado Hospital - Anschutz Cancer Pavillion, Aurora, Colorado
  - Yale University School of Medicine - Department of Neurosurgery, New Haven, Connecticut
  - Florida Hospital Neuroscience Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation, Inc. - Dept of Neurological Surgery, Chicago, Illinois
  - CINN at Rush Unversity Medical School, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - The Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center Department of Neurology, New York, New York
  - Weill Cornell Medical College - Department of Neurological Surgery, New York, New York
  - Columbia University Medical Center - Neurological Institute, New York, New York
  - Carolina Neurosurgery & Spine Assoc., Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences - Department of Neurosurgery, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation Department of Neurological Surgery, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Insitute, Salt Lake City, Utah
  - University of Virginia Health Systems - Department of Neurological Surgery, Charlottesville, Virginia
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington
  - West Virginia University Department of Neurosurgery, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinic, Madison, Wisconsin
- Canada (8):
  - Calgary Health Region, Calgary, Alberta
  - Walter MacKenzie Health Sciences Center, Edmonton, Alberta
  - Cancer Care Manitoba, Winnepeg, Manitoba
  - London Regional Cancer Center, London, Ontario
  - Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Toronto Western Hospital Division of Neurosurgery, Toronto
- Germany (5):
  - Techniche Universität Dresden Klinik und Poliklinik für Neurochirurgie, Dresden
  - Universitätsklinikum Hamburg-Eppendorf - Klinik für Neurochirurgie, Hamburg
  - Klinikum der Universität Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein - Klinik für Neurochirurgie, Kiel
  - Ludwig-Maximilians-Universität München - Klinikum Großhadern - Neurochirurgische Klinik und Poliklinik, München
- Israel (3):
  - Rabin Medical Center - Department of Neurosurgery, Petah Tikva
  - Tel Aviv Sourasky Medical Center (TASMC), Tel Aviv
  - Sheba Medical Center - Department of Neurosurgery, Tel Litwinsky
- Netherlands (2):
  - Academisch Ziekenhuis Groningen Afd. Neurochirurgie, Groningen
  - Erasmus University MC, Rotterdam, Rotterdam
- United Kingdom (2):
  - Institute of Neurological Sciences, Glasgow
  - The Walton Centre for Neurology & Neurosurgery, Liverpool

REFERENCES:
- See also: Click here for more information regarding The PRECISE Trial. — http://www.neophrm.com/index.php?section=1